CLINICAL TRIAL: NCT01862211
Title: POLYGEN DEFI-ALPHA : Genetic Polymorphisms Study in Children With Alpha-1 Antitrypsin Deficiency, Included in the DEFI-ALPHA Cohort
Brief Title: Polygen Defi-Alpha: Genetic Polymorphisms Study in Children With Alpha-1 Antitrypsin Deficiency, Included in the DEFI-ALPHA Cohort
Acronym: Polygen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011.663; ID RCB (Other: 2012-A00204-39.)
Record Dates: First submitted 2013-05-22; First posted 2013-05-24 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Children With a Deficiency of Alpha-1 Antitrypsin
Keywords: alpha antitrypsin, hepatic disease, genetic, polymorphism
MeSH Terms: conditions — Digestive System Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- members of family of children with a DA1AT (Experimental)
  Interventions: Other: blood sampling
- children with a DA1AT (Experimental)
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — A blood sampling will be performed for the genetic analysis and the measurement of serum IL-8.

SUMMARY:
The deficiency of alpha-1 antitrypsin (DA1AT) is a genetic disorder of variable clinical expression, initially described in adults with pulmonary emphysema patients. In children, it is the second cause of neonatal cholestasis after biliary atresia and is a common indication for liver transplantation.

Several genotypes for SERPINA1 gene coding for alpha-1 anti-trypsin were identified. The main ones are M / M, M / Z, M / S and Z / Z and each genotype is closely correlated with the concentration of blood A1AT. The estimate for France suggests a prevalence of genotype deficit Z / Z of the order of 1/6054, (9982 patients), which in 11% of cases, have liver disease (prolonged neonatal jaundice). Half of them will move towards the development of cirrhosis with portal hypertension, at worst liver transplantation.

Currently, we do not know what are the clinical and genetic factors that predispose a patient A1AT deficiency develop liver damage. Recent studies have led us to think that polymorphisms in the gene SERPINA1, as well as that of the alpha-mannosidase 1 endoplasmic reticulum (Erman gene) could be a predictive marker of liver complications. Another possible candidate gene is one of the importin beta (KPNB1), a protein involved in the elimination of misfolded proteins. These data lead us to propose the study of genetic polymorphisms.

The main objective of the study is to compare the allele frequencies of these polymorphisms between (i) a cohort of A1AT deficient patients and with hepatic symptoms (portal hypertension and its complications, severe liver failure leading to transplant or not, or an indication for liver transplantation) and (ii) a cohort of A1AT deficient patients without signs of hepatic call. To build this last cohort, we will include in the genetic study the family members of deficient patients, some of whom probably carrying a deficit genotype Z / Z but without any associated clinical manifestations. This will allow us to facilitate the establishment of genotype profiles / phenotype clearly identified, which then allow a more appropriate care for children who may have such a development, we will strive to achieve a haplotype interpretation of polymorphisms found.

This study will be conducted in association with the DEFI-ALPHA study to identify clinical and biological prognostic factors such as age at diagnosis, the diagnostic mode, the results of liver biopsy (when available), the clinical course, family history, the existence of IUGR and long-term treatment.

The secondary objectives of the study are :

* The measurement and interpretation of serum IL-8 in A1AT-deficient patients. Indeed, one study showed a higher IL-8 in patients with ulcerative colitis compared with healthy patients' serum. These considerations led us to hypothesize that IL-8 may be a marker of liver disease in A1AT deficiency.
* Preservation of blood samples for further study of other genes, which may be in the future suspected to be associated with the occurrence of liver complications. To this end, a DNA bank will be created. It will involve the children with a deficiency of alpha-1 antitrypsin and their family of 1st and 2nd degree in civil law (parents and siblings).

This study is a continuation of the cohort DEFI-ALPHA (descriptive study of a cohort of children with DA1AT) and sought to identify the clinical and biological factors such as age at diagnosis, diagnosis mode, the result sets of the liver biopsy (when available), clinical course, family history, the presence of IUGR and long-term treatment.

The only criterion for not-inclusion is, according to the subject, the lack of consent of the child and his parents, the lack of consent of the adult patient, or the lack of consent of the witness. Demographic and clinical history data (for parents and brothers/sisters showing no DA1AT) will be collected.

Currently, the cohort of patients with DA1AT is being set up in the framework of the "Cohort DEFI-ALPHA." This multicenter project is realized with the help of french pediatric hepatology centers that regularly follow patients DA1AT. Today, over 100 patients DA1AT have already been identified, and the collection of historical data has already begun on several centers since September 2009. This study is therefore a continuation of this work.

Over a period of 30 months, the total number of potentially includable subjects is estimated at about 400 in this study (100 patients and 300 related to the first degree such as parents, brothers and sisters).

This study will be promoted by the Hospices Civils de Lyon. Authorization of the competent authority and the ethical committee will be obtained as well as informed consent from families before blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Children included in the DefiAlpha cohort or adult aged under 18 years at the time of inclusion in the cohort Defi-Alpha, with a deficiency of of alpha-1 antitrypsin
* Beneficiaries subjects of a social security system
* Presence of a signed informed consent (patient or parents) at the time of inclusion

Exclusion Criteria:

- Lack of consent

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2013-05; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
presence of mutations / polymorphisms in genes SERPINA1, Ermani and KPNB1 (with haplotype interpretation) in children with hepatic complications | 1 day
  The main objective of the study is to compare the allele frequencies of these polymorphisms between (i) a cohort of A1AT deficient patients and with hepatic symptoms (portal hypertension and its complications, severe liver failure leading to transplant or not, or an indication for liver transplantation) and (ii) a cohort of A1AT deficient patients without signs of hepatic call.

SECONDARY OUTCOMES:
measurement and interpretation of serum IL-8 | 1 day
  The measurement and interpretation of serum IL-8 in A1AT-deficient patients. Indeed, one study showed a higher IL-8 in patients with ulcerative colitis compared with healthy patients' serum. These considerations led us to hypothesize that IL-8 may be a marker of liver disease in A1AT deficiency.
Identification of modifier genes or mutations responsible of hepatic complications | 1 year
  Find genes responsible of hepatic complications in A1AT-deficient patients by sequencing whole exome

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - CHU d'Amiens - Hopital Nord, Amiens
  - CHU de BESANCON, Besançon
  - Hôpital Pellegrin, Bordeaux
  - Hôpital Femme Mère Enfant de Lyon, Bron
  - CHU Estaing, Clermont-Ferrand
  - Hôpital Couple Enfant, La Tronche
  - CHG Le HAVRE, Le Havre
  - AP-HP - Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Jeanne de Flandre, Lille
  - Hopital de la Timone, Marseille
  - Hôpital Brabois Enfants, Nancy
  - Hôpital Mère Enfant, Nantes
  - AP-HP Hôpital Necker, Paris
  - Hôpital Anne de Bretagne, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Hôpital Nord, Saint-Etienne
  - CH Saint Nazaire, Saint-Nazaire
  - Hopital Hautepierre, Strasbourg
  - Hôpital des Enfants, Toulouse
  - Centre de Pédiatrie Gatien de Clocheville, Tours

REFERENCES:
- [Background] Ruiz M, Lacaille F, Berthiller J, Joly P, Dumortier J, Aumar M, Bridoux-Henno L, Jacquemin E, Lamireau T, Broue P, Rivet C, Belmalih A, Restier L, Chapuis-Cellier C, Bouchecareilh M, Lachaux A; Groupe Francophone d'Hepatologie Gastroenterologie et Nutrition Pediatriques. Liver disease related to alpha1-antitrypsin deficiency in French children: The DEFI-ALPHA cohort. Liver Int. 2019 Jun;39(6):1136-1146. doi: 10.1111/liv.14035. Epub 2019 Feb 1. PMID 30589493
- [Result] Joly P, Ruiz M, Garin R, Karatas E, Lachaux A, Restier L, Belmalih A, Renoux C, Lombard C, Dechomet M, Bouchecareilh M. A Particular SORL1 Micro-haplotype May Prevent Severe Liver Disease in a French Cohort of Alpha 1-Antitrypsin-deficient Children. J Pediatr Gastroenterol Nutr. 2021 Sep 1;73(3):e68-e72. doi: 10.1097/MPG.0000000000003125. PMID 33720088